CLINICAL TRIAL: NCT04491617
Title: STandard Versus No Opioid Prescription After Prolapse and Anti-INcontinence Surgery: A Randomized Controlled, Non-inferiority Trial
Brief Title: STandard Versus No Opioid Prescription After Prolapse and Anti-INcontinence Surgery Trial
Acronym: STOP-PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-682
Record Dates: First submitted 2020-07-08; First posted 2020-07-29 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain; Opioid Use; Prolapse; Female; Incontinence
Keywords: Opioids; Gynecology; Pain control; Prolapse; Incontinence
MeSH Terms: conditions — Pain, Postoperative; Prolapse; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Opioid Protocol (Control) (Active Comparator): Standard postoperative medications (opioids and non-opioids) are prescribed upon discharge after surgery
  Interventions: Other: Standard opioid prescribing
- Restrictive Opioid Protocol (Intervention) (Experimental): Only non-opioid analgesics (i.e. ibuprofen and acetaminophen) are prescribed upon discharge after surgery. Patients are allowed to request an opioid prescription if they so desire
  Interventions: Other: Restrictive opioid prescribing

INTERVENTIONS:
Other: Standard opioid prescribing — Patients are routinely prescribed opioid medications in addition to non-opioids.
  Arms: Standard Opioid Protocol (Control)
Other: Restrictive opioid prescribing — Patients are prescribed non-opioid pain medications, and will be prescribed opioids only if they request them.
  Arms: Restrictive Opioid Protocol (Intervention)

SUMMARY:
Overprescribing opioids is considered a major contributor to the opioid crisis. Hill et al. demonstrated that within a general surgery practice, over 70% of the prescribed opioid pills were never taken. Disturbingly, 45% of patients who did not take opioids at all on their day of discharge were discharged with an opioid prescription (Chen et al). Recent initiatives have attempted to utilize restrictive opioid prescribing protocols for postoperative pain management in which patients were prescribed a limited number of opioid tablets (Hallway et al) or prescribed opioids only if they were used as an inpatient (Mark et al). These well-conducted studies show that restrictive opioid prescribing policies achieve the goal of reducing excess opioid exposure without causing undue harm, inconvenience or dissatisfaction among patients.

The objective of this study is to determine if a restrictive opioid prescription protocol (in which patients are not prescribed postoperative opioids unless they request them) is acceptable to patients after ambulatory and major urogynecologic surgery, compared to standard opioid prescribing practices. The study investigators believe that physicians can capitalize on the new ability to electronically prescribe opioids for patients who require them, to prevent over-prescribing without impacting patient care. The study also intends to describe postoperative opioid use patterns in the urogynecologic population, including factors predictive of opioid use and non-use. The results of this research will have a significant and timely impact by helping to reduce opioid overprescribing and informing future prescribing guidelines in the field of urogynecology.

DETAILED DESCRIPTION:
Specific Aims

Aim 1. To compare patient satisfaction and pain control using two different opioid prescribing protocols.

The study investigators hypothesize that postoperative pain control and satisfaction will be non-inferior between patients not routinely prescribed opioids after surgery and those prescribed a standard quantity. Participants will be asked to rate their pain control during the first 7 postoperative days with validated questionnaires. Participants' satisfaction with pain control will be evaluated at their postoperative visit.

Aim 2. To examine opioid use patterns after ambulatory and major urogynecologic surgery.

The study investigators hypothesize that most postoperative patients will use few or no opioids after urogynecologic surgery, regardless of prescribing protocol. All participants will receive thorough counseling with detailed instructions on non-opioid pain management, as well as multimodal analgesia via ERAS protocol during the perioperative period. Participants will be asked to log their opioid and non-opioid medication use in the first postoperative week. The investigators will also assess the number of requests for opioid prescription (in those randomized to the restrictive protocol) and opioid refills (from patients in the standard protocol).

Aim 3. To determine patient and perioperative factors associated with opioid use after urogynecologic surgery.

The study investigators plan to collect and analyze demographic, clinical and psychometric data on all participants with the goal of predicting analgesic needs and opioid use after urogynecologic surgery. Results from this study will guide surgeons on how to tailor opioid prescriptions to the needs of each patient, based off individual patient and perioperative characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* Access to ancillary care, including phone advice, nurse and outpatient clinic numbers
* Transportation to outpatient clinic or ability to access Virtual Care Visits
* Able to speak and read English
* Has decision-making capacity and able to provide consent for research participation

Exclusion Criteria:

* History of substance abuse disorder
* Chronic opioid use
* Score greater than or equal to 30 on Pain Catastrophizing Scale
* Allergy (not intolerance) to greater than or equal to 2 opioids
* Contraindications to both NSAIDs and acetaminophen
* Surgery scheduled on Friday or before major federal holiday
* Patients undergoing concomitant colorectal procedures
* Patients with perioperative complication (such as iatrogenic bowel and bladder injury, hemorrhage, unanticipated laparotomy or ICU admission)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Ferrando, M.D., M.P.H., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Chen EY, Marcantonio A, Tornetta P 3rd. Correlation Between 24-Hour Predischarge Opioid Use and Amount of Opioids Prescribed at Hospital Discharge. JAMA Surg. 2018 Feb 21;153(2):e174859. doi: 10.1001/jamasurg.2017.4859. Epub 2018 Feb 21. PMID 29238810
- [Background] Hallway A, Vu J, Lee J, Palazzolo W, Waljee J, Brummett C, Englesbe M, Howard R. Patient Satisfaction and Pain Control Using an Opioid-Sparing Postoperative Pathway. J Am Coll Surg. 2019 Sep;229(3):316-322. doi: 10.1016/j.jamcollsurg.2019.04.020. Epub 2019 May 30. PMID 31154092
- [Background] Mark J, Argentieri DM, Gutierrez CA, Morrell K, Eng K, Hutson AD, Mayor P, Szender JB, Starbuck K, Lynam S, Blum B, Akers S, Lele S, Paragh G, Odunsi K, de Leon-Casasola O, Frederick PJ, Zsiros E. Ultrarestrictive Opioid Prescription Protocol for Pain Management After Gynecologic and Abdominal Surgery. JAMA Netw Open. 2018 Dec 7;1(8):e185452. doi: 10.1001/jamanetworkopen.2018.5452. PMID 30646274
- [Background] Davidson ERW, Paraiso MFR, Walters MD, Propst K, Ridgeway B, Yao M, Ferrando CA. A randomized controlled noninferiority trial of reduced vs routine opioid prescription after prolapse repair. Am J Obstet Gynecol. 2020 Oct;223(4):547.e1-547.e12. doi: 10.1016/j.ajog.2020.03.017. Epub 2020 Mar 19. PMID 32199926
- [Background] Barber MD, Janz N, Kenton K, Hsu Y, Greer WJ, Dyer K, White A, Meikle S, Ye W. Validation of the surgical pain scales in women undergoing pelvic reconstructive surgery. Female Pelvic Med Reconstr Surg. 2012 Jul-Aug;18(4):198-204. doi: 10.1097/SPV.0b013e31825d65aa. PMID 22777367
- [Derived] Yuan AS, Propst KA, Ross JH, Wallace SL, Paraiso MFR, Park AJ, Chapman GC, Ferrando CA. Restrictive opioid prescribing after surgery for prolapse and incontinence: a randomized, noninferiority trial. Am J Obstet Gynecol. 2024 Mar;230(3):340.e1-340.e13. doi: 10.1016/j.ajog.2023.10.027. Epub 2023 Oct 18. PMID 37863158

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
Started | 64 | 65
Completed | 64 | 63
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention) | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 92
  >=65 years | 19 | 16 | 35
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [31 to 85] | 55.9 [26 to 73] | 56.3 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 59 | 63 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Satisfied With Pain Control at 6 Week Postoperative Visit
Description: The proportion of patients satisfied with postoperative pain control will be reported. Patient satisfaction with pain control was assessed with a 5-point Likert scale at the postoperative visit ("Overall, how satisfied were you with your postoperative pain medication?" [ranked 1- Very Dissatisfied to 5- Very Satisfied] and those who ranked their satisfaction level as a 4 or 5 were considered satisfied.
Time Frame: 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
Number analyzed (Participants) | 64 | 63
Participants | 59 | 58

2. Secondary Outcome: Pain Level Scores During First Postoperative Week
Description: Patients will be asked to report their pain level for the first 7 days postoperatively. Pain levels will be assessed using questions 1, 2 and 4 from the Modified Surgical Pain Scales (SPS), which measures pain at rest, during normal activities and quantifies unpleasantness of worst pain using an 11-point numeric rating score, with 0 representing 'No pain sensation' and 10 representing 'Most intense pain imaginable'. Higher scores indicate a greater amount of pain. REDCap or paper surveys will be used.
Time Frame: 1-week
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
Number analyzed (Participants) | 64 | 65
score on a scale
  Day 1 | 7 [4 to 8] | 6 [3 to 8]
  Day 2 | 6 [3 to 8] | 5 [3 to 8]
  Day 3 | 5 [3 to 7] | 4 [2 to 7]
  Day 4 | 4 [2 to 6] | 4 [2 to 6]
  Day 5 | 3 [2 to 6] | 3 [2 to 6]
  Day 6 | 3 [1 to 5] | 3 [1 to 4]
  Day 7 | 2 [1 to 4] | 2 [1 to 4]

3. Secondary Outcome: Opioid Usage in the First Postoperative Week
Description: Participants will be asked to log opioid and non-opioid medication in number of tablets used during the first postoperative week with either REDCap or paper surveys. The opioid usage by study arm was reported in mean morphine equivalents (MMEs).
Time Frame: 1-week
Measure: Median (Inter-Quartile Range); unit: MMEs
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
Number analyzed (Participants) | 64 | 65
MMEs | 0 [0 to 15] | 0 [0 to 8]

4. Secondary Outcome: Number of Participants Who Requested a New Opioid Prescription or Opioid Refill
Description: Investigators will track the number of participants who requested a new opioid prescription or opioid refill during the 6 week postoperative period.
Time Frame: 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
Number analyzed (Participants) | 64 | 30
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Standard Opioid Protocol (Control) | Restrictive Opioid Protocol (Intervention)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/63
Other Adverse Events (participants affected / at risk) | 0/64 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04491617/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT04491617/ICF_001.pdf